CLINICAL TRIAL: NCT04434001
Title: ZEPLAST- PED: ZEro_PLASma Trial in Small Infants Undergoing Cardiac Surgery Randomized Controlled Pilot Phase II Study
Brief Title: ZEPLAST- PED: ZEro_PLASma Trial in Small Infants Undergoing Cardiac Surgery
Acronym: ZEPLAST-PED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study encountered unexpected difficulties in enrolling patients due to requirements for the Informed Consent. 60% of our patients comes from abroad with only one accompanying parent. The rules of our EC require both parents to sign the consent.
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Head of Cardiothoracic and Vascular Anesthesia and Intensive Care, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZEPLAST-PED
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Bleeding; Cardiac Defect; Surgery--Complications; Fibrinogenopenia; Acquired; Transfusion-Related Acute Lung Injury; Transfusion-Associated Circulatory Overload; Congenital Heart Disease
Keywords: bleeding; pediatric cardiac surgery; fresh frozen plasma; fibrinogen concentrate; prothrombin complex concentrate
MeSH Terms: conditions — Hemorrhage; Afibrinogenemia; Transfusion-Related Acute Lung Injury; Transfusion Reaction; Heart Defects, Congenital; Hemophilia B | interventions — Fibrinogen; Factor IX

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZEPLAST (Experimental): In case of bleeding and:
  * CT INTEM > CT HEPTEM by 25% : give protamine 0.25 mg/kg;
  * MCF FIBTEM < 8 mm : give Fibrinogen Concentrate 30 mg/kg;
  * CT EXTEM > 100 s : give Prothrombin Complex Concentrate 20 mg/kg.
  Interventions: Drug: Fibrinogen Concentrate Human; Drug: Prothrombin Complex Concentrate
- Control (Active Comparator): In case of bleeding and:
  * CT INTEM > CT HEPTEM by 25% : give protamine 0.25 mg/kg;
  * fibrinogen and/or thrombin generation deficiency : give FFP 10-20 ml/kg.
  Interventions: Biological: Fresh Frozen Plasma

INTERVENTIONS:
Drug: Fibrinogen Concentrate Human — Treatment of acquired postoperatively fibrinogen deficiency as assessed by ROTEM FIBTEM test.
  Other Names: Haemocomplettan
  Arms: ZEPLAST
Drug: Prothrombin Complex Concentrate — Treatment of acquired postoperatively thrombin generation deficiency as assessed by ROTEM EXTEM test.
  Other Names: Confidex
  Arms: ZEPLAST
Biological: Fresh Frozen Plasma — Treatment of acquired postoperative coagulopathy as assessed by ROTEM FIBTEM and INTEM tests.
  Arms: Control

SUMMARY:
In pediatric patients (newborns and infants weighing less than 10 kg) undergoing cardiac surgery with extracorporeal circulation postoperative bleeding represents a known complication with a significant impact on outcome. Fresh frozen plasma (FFP) for bleeding management is associated, particularly in this kind of patients, to volume overload and a significative increase of Transfusion Related Acute Lung Injury (TRALI), further worsening the postoperative outcome. In the adult patient FFP employment could be almost completely canceled by administration of concentrated hemostatic components - the fibrinogen concentrate and prothrombin complex concentrate (PCC). We designed this phase II pilot study to establish whether an analogous strategy, modified accordingly to pediatric physiology, could be safely and successfully applied in newborns and infants.

DETAILED DESCRIPTION:
The study population will be randomized to two groups: ZEPLAST and control, respectively.

The two groups will receive the same priming solution (containing Red Blood Cells and albumin 5%) and heparin/protamine management. In both groups coagulation will be assessed with rotational thromboelastometry (ROTEM - EXTEM, INTEM, HEPTEM and FIBTEM tests) after heparin antagonization. In case of bleeding, coagulopathies will be treated differently:

* in the ZEPLAST group, fibrinogen deficiency (FIBTEM Maximum Clot Firmness MCF < 8 mm) will be treated with 30 mg/kg of concentrated fibrinogen; low thrombin generation (EXTEM Clotting Time CT > 100 s) will be treated with 20 mg/kg of prothrombin complex concentrate;
* in the control group, coagulopathies will be treated with 10-20 ml/kg of FFP. In case of refractory bleeding, PCC and fibrinogen can be administered as a rescue treatment.

Further ROTEM tests will be performed at 24 and 48 hours post surgery. Outcome parameters will be collected at the same timepoints.

ELIGIBILITY:
Inclusion Criteria:

* newborns and infants with weight lower than 10 kg undergoing cardiac surgery with extracorporeal circulation:
* informed consent signed by both parents or legal guardian.

Exclusion Criteria:

* emergency surgery;
* known congenital coagulopathy or suspected based on anamnesis;
* participation to other clinical trials;
* known hypersensitivity to components and excipients of FFP , prothrombin complex concentrate or fibrinogen concentrate.

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Transfusion of Fresh Frozen Plasma (FFP) | First 48 hours after surgery
  Number of patients transfused with FFP

SECONDARY OUTCOMES:
Postoperative bleeding | First 12, 24 and 48 hours after surgery
  Amount of blood collected by chest drainages
Severe bleeding | First 12 hours after surgery
  Number of patients who experienced severe bleeding (higher than 30 ml/kg in the first 12 hours after surgery)
Surgical re-exploration for bleeding | First 12, 24 and 48 hours after surgery
  Number of patients requiring surgical re-exploration due to bleeding (bleeding with no coagulopathies detected or refractory to pharmacological treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore SB. Transfusion-related acute lung injury (TRALI): clinical presentation, treatment, and prognosis. Crit Care Med. 2006 May;34(5 Suppl):S114-7. doi: 10.1097/01.CCM.0000214312.20718.3E. PMID 16617254
- [Background] Ranucci M, Baryshnikova E. Fibrinogen supplementation after cardiac surgery: insights from the Zero-Plasma trial (ZEPLAST). Br J Anaesth. 2016 May;116(5):618-23. doi: 10.1093/bja/aev539. Epub 2016 Feb 17. PMID 26893405
- [Background] Bianchi P, Cotza M, Beccaris C, Silvetti S, Isgro G, Pome G, Giamberti A, Ranucci M; Surgical and Clinical Outcome REsearch (SCORE) group. Early or late fresh frozen plasma administration in newborns and small infants undergoing cardiac surgery: the APPEAR randomized trial. Br J Anaesth. 2017 May 1;118(5):788-796. doi: 10.1093/bja/aex069. PMID 28510741
- [Background] Ranucci M, Bianchi P, Cotza M, Beccaris C, Silvetti S, Isgro G, Giamberti A, Baryshnikova E. Fibrinogen levels and postoperative chest drain blood loss in low-weight (<10 kg) children undergoing cardiac surgery. Perfusion. 2019 Nov;34(8):629-636. doi: 10.1177/0267659119854246. Epub 2019 Jun 28. PMID 31250738
- [Derived] Hayes K, Fernando MC, Jordan V. Prothrombin complex concentrate in cardiac surgery for the treatment of coagulopathic bleeding. Cochrane Database Syst Rev. 2022 Nov 21;11(11):CD013551. doi: 10.1002/14651858.CD013551.pub2. PMID 36408876